CLINICAL TRIAL: NCT02985788
Title: Validation of Self Digital Photography for Assessing Elbow Range of Motion
Brief Title: Self Digital Photography for Assessing Elbow Range of Motion
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shawn W. O'Driscoll, PI, Mayo Clinic
Other Study IDs: 13-003378
Record Dates: First submitted 2016-11-08; First posted 2016-12-07 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Contracture of Elbow Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Video Instructions: Instructions on how to take a flexion/extension picture will be delivered in video format. These instructions will be followed by written instruction on how to take pictures examining pronation/supination.
- Written instructions: Instructions on how to take a flexion/extension picture will be delivered in a written, on paper format. These instructions will be followed by written instruction on how to take pictures examining pronation/supination.

SUMMARY:
Loss of elbow range of motion can significantly affect activities of daily living. Measuring elbow range of motion is critical for tracking post surgical outcomes. This study seeks to validate the ability to validate self photography as a means of followup through long distance correspondence.

DETAILED DESCRIPTION:
Loss of elbow range of motion is common after trauma and can significantly affect activities of daily living. Patients across the country travel to tertiary referral centers to have this problem addressed. Followup is critical and can often be difficult given distances between patients home and their healthcare provider. Measuring postoperative outcomes requires accurate and reliable documentation of range of motion. Previously, the investigators have validated digital photography as a means of accurately measuring elbow range of motion. In that study, photographs were taken by a non-professional photographer. With the advance in personal technology, patients now have the ability to take photos themselves. This study seeks to validate self photography, which will ultimately improve patient follow up and improve clinical monitoring

ELIGIBILITY:
Inclusion Criteria:

* Elbow contracture in the sagittal place

Exclusion Criteria:

* Unable to read English
* Unable to forward flex shoulder to 90 degrees or hold their shoulder at 90 degrees for the duration of the examination
* Unable to tolerate the exercise due to pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have an elbow contracture in the sagittal plane
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Digital photo-based elbow range of motion measurement compared to traditional goniometry | up to 2 months
  Patients will follow instructions to take a photograph of themselves capturing elbow range of motion (flexion, extension, supination and pronation). Elbow range of motion will then be measured clinically with a goniometer. Patient's active participation will be 1 day. Range of motion will be measured off of photographs 1 month after capturing pictures and repeated 2 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Shawn O'Driscoll, PhD MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided